CLINICAL TRIAL: NCT02607033
Title: Exercise and Weight Loss to Improve Mobility Function in Veterans With PAD
Brief Title: Exercise and Weight Loss in PAD
Acronym: Action3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1788-W; IK2RX001788-01 (NIH)
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Exercise; Weight Loss; Mobility Limitation
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Weight Loss; Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and Weight Loss (Experimental): Individuals assigned to this group will be asked to complete both the exercise and weight loss intervention for six months
  Interventions: Other: Exercise; Other: Weight Loss
- Exercise (Active Comparator): Individuals assigned to this group will be asked to complete the exercise intervention for xic months
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Individuals will be asked to walk 3 times a week on a treadmill (initially starting at 15 minutes and progressing up to 40 minutes) and participate in a short weight training program focused on increasing strength in the legs.
Other: Weight Loss — Individuals will be asked to meet with a registered dietitian once a week to discuss strategies to reduce daily caloric intake to gradually reduce body weight over 6 months.
  Arms: Exercise and Weight Loss

SUMMARY:
This study is designed to examine the added benefits of weight loss to an exercise program in older obese Veterans with peripheral arterial disease. The investigators want to determine if weight loss in addition to exercise will 1) improve walking ability to a greater extent than exercise alone and 2) determine the underlying reasons why walking ability improves by measuring blood flow and the amount of muscle in the leg muscles.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects an estimated 12 -15 million adults in the US and an estimated 20% of older Veterans. Those with PAD ambulate with slow gait and experience decreased leg strength, dysmobility, reduced quality of life, serious morbidity and often premature death. It is estimated that over 60% of individuals with PAD are overweight or obese. While PAD itself worsens mobility, obesity adds a further functional burden to older adults with PAD. Individuals diagnosed with PAD, who are also obese typically claudicate 40% more quickly than non-obese individuals and take 20% longer to recover after claudication. Studies of older obese adults without PAD have demonstrated that the combination of exercise and weight loss is more effective at improving physical function and body composition than exercise alone. While these findings likely translate to older adults with PAD, this hypothesis has yet to be tested. This study is designed to determine whether weight loss and exercise (WL+EX) versus exercise ( EX ) alone will 1) improve mobility function (walking ability) to a greater extent than exercise alone and 2) determine the mechanisms underlying changes in mobility function by measuring muscle microvascular perfusion and composition. The investigators hypothesize that a combined intervention of weight loss and exercise (aerobic and restive) will result in greater improvements in mobility function through improved muscle perfusion and reduced muscle fat infiltration than exercise alone in obese Veterans with PAD.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 kg/m2
* Ankle Brachial Index (ABI) <.90
* Able to participate in a supervised exercise program at the Baltimore VA
* No current plan for surgical revascularization
* Claudication or leg symptoms when walking

Exclusion Criteria:

* Unstable angina or a recent heart attack
* Active cancer
* Dementia
* Current foot or leg ulcers
* Already exercise 2x/week or more.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odessa R. Addison, PhD DPT, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise and Weight Loss | Exercise
Started | 9 | 9
Completed | 7 | 2
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise and Weight Loss | Exercise | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 5 | 8 | 13
Age, Continuous [Median (Full Range); unit: years] | 66 [60 to 77] | 72 [58 to 86] | 67 [58 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Difference in Time to Onset of Calf Pain (Claudication Onset Time) Pre-intervention to Post-intervention
Description: The change in the amount of time it takes for calf pain to first appear while walking on a treadmill comparing pre and post-intervention
Time Frame: 6 months
Population: 6 individuals in the exercise and weight loss group and 2 individuals in the exercise group completed pre/post measures for Claudication onset time
Measure: Median (Full Range); unit: seconds
Arm/Group | Exercise and Weight Loss | Exercise
Number analyzed (Participants) | 6 | 2
seconds | 396 [264 to 524] | 140 [106 to 175]
Statistical Analysis 1: Comparison: Exercise and Weight Loss; Wilxocon signed Rank test to compare pre to post onset of pain time in the Exercise + Weight loss group. Due to low sample size were unable to compare changes between the Exercise + Weight Loss group and the Exercise only groups; Test type: Other — Wilxocon signed Rank test; p = 0.028, Wilxocon signed Rank test

2. Primary Outcome: Difference in Ankle Brachial Index Pre-intervention to Post-intervention
Description: A change in the muscle blood flow to the legs determined by taking blood pressure in the arms and legs before and after cessation of exercise comparing the change pre to post exercise scores pre-intervention (baseline) and post intervention (6 months). There are no units because the ankle brachial index is a ratio. An improvement would be a higher number a post-intervention testing than pre-intervention testing. A negative number indicates improvement while a positive number indicates a worse score post-testing.
Time Frame: 6 months
Population: 6 individuals in the exercise and weight loss group and 2 individuals in the exercise group completed pre/post measures for ankle brachial index
Measure: Median (Full Range); unit: ratio
Arm/Group | Exercise and Weight Loss | Exercise
Number analyzed (Participants) | 6 | 2
ratio | 0.04 [-0.15 to 0.27] | -0.16 [-0.18 to -0.14]

3. Secondary Outcome: Score on the Modified Physical Performance Test Post-intervention
Description: A mobility measure that utilizes 9 tasks scored 0-4 (total possible score 36) to determine functional status. Scores from each of the nine items are summed for the total score. Scores are from 0-36 with higher scores considered to be better. The post-testing median score will be reported for post-testing.
Time Frame: 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Exercise and Weight Loss | Exercise
Number analyzed (Participants) | 7 | 2
score on a scale | 33 [30 to 36] | 31 [26 to 36]

4. Secondary Outcome: Change in Muscle Composition of the Calf Muscles Pre-intervention to Post-intervention
Description: A measure of the amount of muscle and fat in the muscle using a CT scan of the legs. Pre-test levels will be compared to post-test levels.
Time Frame: 6 months
Population: This measure was not conducted due to staffing and pandemic related limitations in acquiring the CT scans.
Arm/Group | Exercise and Weight Loss | Exercise
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months from baseline
Arm/Group | Exercise and Weight Loss | Exercise
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9 | 3/9
Other Adverse Events (participants affected / at risk) | 4/9 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise and Weight Loss (N=9) | Exercise (N=9)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — New onset of Cerebrovascular accident (CVA)
angina (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Bypass Graft (CABG) (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal (GI) bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise and Weight Loss (N=9) | Exercise (N=9)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (5) | 2 (3)
Car accident (Social circumstances) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Lower recruitment with an overall small sample size limited the number of participants to be analyzed in the study. An unequal drop out rate between the groups also limits interpretation of data at the six-month time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT02607033/Prot_SAP_000.pdf